CLINICAL TRIAL: NCT03676322
Title: A Phase I, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses and Multiple Ascending Doses of M5049 Administered Orally in Healthy Participants
Brief Title: Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) Study of M5049 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MS200569_0001; 2018-001256-35 (EudraCT Number)
Record Dates: First submitted 2018-09-17; First posted 2018-09-18 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Healthy
Keywords: Pharmacokinetics; M5049

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Part A: M5049 (Experimental)
  Interventions: Drug: M5049
- Part A: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Part B: M5049 (Experimental)
  Interventions: Drug: M5049
- Part B: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Part C: M5049 (Experimental)
  Interventions: Drug: M5049

INTERVENTIONS:
Drug: M5049 — Participants will receive single ascending oral dose of M5049 in Part A. Participants will receive multiple ascending oral dose of M5049 once daily for 14 days or twice daily for 13 days followed by a single dose on Day 14 in the morning in Part B. Participants will receive a single oral dose of M5049 under fed conditions in Part C.
  Arms: Part A: M5049; Part B: M5049; Part C: M5049
Drug: Placebo — Participants will receive placebo matched to M5049.
  Arms: Part A: Placebo; Part B: Placebo

SUMMARY:
The study will evaluate the safety, tolerability, Pharmacokinetic (PK), Pharmacodynamics (PD), and explore the food effect of M5049 in healthy male and female participants.

ELIGIBILITY:
Inclusion Criteria:

* Body weight between 50 to 100 kilogram (kg)
* Body mass index (BMI) between 18.5 and 29.9 kilogram per meter square (kg/m^2)
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* History of clinically relevant disease of any organ system that may interfere with the objectives of the study or provide a risk to the health of the participant
* History of splenectomy
* History of epilepsy, other neurological disorders, or neuropsychiatric conditions
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2019-07-26 (Actual); Study Completion 2019-07-26 (Actual)

PRIMARY OUTCOMES:
Part A: Occurrence and Severity of Treatment-emergent Adverse Events (TEAEs) and Serious AEs (SAEs) | Day 1 up to Day 21
Part A: Number of Participants With Clinically Significant Changes in Vital Signs, Laboratory Parameters and 12-lead Electrocardiogram (ECG) Findings | Day 1 up to Day 21
  Number of participants with clinically significant changes will be reported.
Part B: Occurrence and Severity of TEAEs and SAEs | Day 1 up to Day 33
Part B: Number of Participants With Clinically Significant Changes in Vital Signs, Laboratory Parameters and 12-lead Electrocardiogram (ECG) Findings | Day 1 up to Day 33
  Number of participants with clinically significant changes will be reported.
Part C: Maximum Observed Plasma Concentration (Cmax) of M5049 | Pre-dose up to Day 6
Part C: Time to Reach Maximum Plasma Concentration (tmax) of M5049 | Pre-dose up to Day 6
Part C: Elimination Rate Constant (λz) of M5049 | Pre-dose up to Day 6
Part C: Apparent Terminal Half-life (t1/2) of M5049 | Pre-dose up to Day 6
Part C: Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Sampling Time (AUC 0-t) of M5049 | Pre-dose up to Day 6
Part C: Area Under the Concentration-Time Curve Over Entire Dosing Time Period From Time Zero Extrapolated to Infinity (AUC0-inf) | Pre-dose up to Day 6
Part C: Total Body Clearance (CL/f) of M5049 | Pre-dose up to Day 6
Part C: Apparent Volume of Distribution (Vz/f) of M5049 | Pre-dose up to Day 6

SECONDARY OUTCOMES:
Part A: Maximum Observed Blood Concentration (Cmax) of M5049 | Pre-dose up to Day 6
Part A: Time to Reach Maximum Plasma Concentration (tmax) of M5049 | Pre-dose up to Day 6
Part A: Elimination Rate Constant (λz) of M5049 | Pre-dose up to Day 6
Part A: Apparent Terminal Half-life (t1/2) of M5049 | Pre-dose up to Day 6
Part A: Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Sampling Time (AUC 0-t) of M5049 | Pre-dose up to Day 6
Part A: Area Under the Concentration-Time Curve Over Entire Dosing Time Period From Time Zero Extrapolated to Infinity (AUC0-inf) | Pre-dose up to Day 6
Part A: Total Body Clearance (CL/f) of M5049 | Pre-dose up to Day 6
Part A: Apparent Volume of Distribution (Vz/f) of M5049 | Pre-dose up to Day 6
Part A: Dose Normalized Maximum Observed Plasma Concentration (Cmax/D) of M5049 | Pre-dose up to Day 6
Part A: Dose Normalized Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Sampling Time (AUC0-t/D) of M5049 | Pre-dose up to Day 6
Part A: Change From Baseline in QT Interval Corrected Using Fridericia's Formula (QTcF) on Digital Holter Electrocardiograms (ECG) at Day 2 | Baseline, Day 2
Part A: Time Matched Plasma Concentration of M5049 | Pre-dose up to Day 6
Part B: Maximum Observed Blood Concentration (Cmax) of M5049 | Pre-dose up to Day 19
Part B: Time to Reach Maximum Plasma Concentration (tmax) of M5049 | Pre-dose up to Day 19
Part B: Elimination Rate Constant (λz) of M5049 | Pre-dose up to Day 19
Part B: Apparent Terminal Half-life (t1/2) of M5049 | Pre-dose up to Day 19
Part B: Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Sampling Time (AUC 0-t) of M5049 | Pre-dose up to Day 19
Part B: Area Under the Concentration-Time Curve Over Entire Dosing Time Period From Time Zero Extrapolated to Infinity (AUC0-inf) | Pre-dose up to Day 19
Part B: Total Body Clearance (CL/f) of M5049 | Pre-dose up to Day 19
Part B: Apparent Volume of Distribution (Vz/f) of M5049 | Pre-dose up to Day 19
Part B: Area Under the Concentration-Time Curve Over the Dosing Interval (AUCtau) | Pre-dose up to Day 19
Part B: Accumulation Ratio for Cmax (Racc Cmax) of M5049 | Pre-dose up to Day 19
Part B: Accumulation Ratio for AUCtau(Racc AUCtau) of M5049 | Pre-dose up to Day 19
Part B: Peak trough Ratio of M5049 | Pre-dose up to Day 19
Part B: Plasma Concentration Prior to the Next Dose (C trough) of M5049 | Pre-dose up to Day 19
Part B: Dose Normalized Maximum Observed Plasma Concentration at Steady State (Cmaxss/D) of M5049 | Pre-dose up to Day 19
Part B: Dose Normalized Area Under the Concentration-Time Curve Over the Dosing Interval (AUCtau/D) of M5049 | Pre-dose up to Day 19
Part B: Change From Baseline in QT Interval Corrected Using Fridericia's Formula (QTcF) on Digital Holter Electrocardiograms (ECG) at Day 2 | Baseline, Day 2
Part B: Time Matched Plasma Concentration of M5049 | Pre-dose up to Day 19
Part C: Occurrence and Severity of Treatment-emergent Adverse Events (TEAEs) and Serious AEs (SAEs) | Day 1 up to Day 23
Part C: Number of Participants With Clinically Significant Changes in Vital Signs, Laboratory Parameters and 12-lead Electrocardiogram (ECG) Findings | Day 1 up to Day 23
  Number of participants with clinically significant changes will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany